## EFFECTS OF METFORMIN AND COMBINATION OF METFORMIN AND PIOGLITAZONE ON PLASMA IL-6 AND IL-8 LEVELS IN POLYCYSTIC OVARIAN SYNDROME

Clinical trial registration number: NCT03117517

Date: 15/03/2018

## Statistical analysis:

The normality of the data was tested using Kolmogorov-Smirinov and Shapiro-Wilk tests and histograms. FSH, LH, Prolactin, testosterone, IL-6 and IL-8 were not normally distributed and were log transformed for analysis. In the final results log transformed values were back transformed and presented as geometric means and confidence intervals. Patient demographic data were evaluated at baseline as descriptive statistics and presented as mean  $\pm$  SD. Wilcoxon signed rank test was used to analyze and compare number of follicles in right and left ovary in the two groups, and also between baseline and follow-up. Results were presented as Median (interquartile range). The baseline data of anthropometric, hormonal and inflammatory markers were compared between the two groups by independent sample t test. Comparison between baseline and after intervention (of 12 weeks) data was done by paired sample t-test for both groups independently. Post intervention comparison between the two groups was also done by independent sample t-test. The change taking place between baseline and after 12 weeks due to intervention was calculated as difference or  $\Delta$ .  $\Delta$  was calculated as value at 12 weeks – value at baseline for hormonal, inflammatory and ovarian size variables. The  $\Delta$  between the two groups was compared by independent sample t-test. P < 0.05 was considered statistically significant. All analyses were performed using SPSS software, version 21 "SPSS (IBM, Armonk, NY, USA).